CLINICAL TRIAL: NCT02628379
Title: A Prospective Observational Trial Evaluating Outcomes of FoundationOne - Directed Matched Targeted Therapy in Patients With Cancer of Unknown Primary (CUP)
Brief Title: Outcomes of FoundationOne Directed Therapy in Cancer of Unknown Primary
Status: Completed | Type: Observational
Sponsor: Foundation Medicine (Industry)
Collaborators: Rush University Medical Center (Other); Stormont-Vail Healthcare (Unknown); Jefferson Medical College of Thomas Jefferson University (Other); The Cleveland Clinic (Other); Sparrow Health System (Other); Cancer & Hematology Centers of Western Michigan (CHCWM) (Unknown); Allegheny Health Network (Other); St. Luke's Hospital and Health Network, Pennsylvania (Other); Solano Hematology Oncology (Unknown); Horizon Oncology Center (Unknown); Comprehensive Blood and Cancer Center (Other); Lancaster Cancer Center (Other); Western Maryland Health Center (Unknown); Valley Medical Oncology (Unknown); Cape Fear Valley Health System (Other); Tri-County Hematology Oncology (Unknown); Hematology & Oncology Associates (Unknown); Broome Oncology (Unknown); Orchard Healthcare (Unknown); Ashland Bellefonte Cancer Center (Unknown); Tennessee Cancer Specialists (Unknown); North Shore Hematology Oncology (Unknown); Good Samaritan (Unknown); Zangmeister Cancer Center (Unknown); Watson clinic (Unknown); Oncology Consultants (Unknown); Oncology Hematology Care (Unknown); Northern Westchester Hospital (Other); Peter MacCallum Cancer Center Trials Unit (Unknown)
Responsible Party: Sponsor
Other Study IDs: RAP-CLT-15-010
Record Dates: First submitted 2015-12-01; First posted 2015-12-11 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Neoplasms, Unknown Primary; CUP; Metastatic Disease; Poorly Differentiated Adenocarcinoma; Poorly Differentiated Carcinoma; Squamous Carcinoma Poorly Differentiated
Keywords: Genomic Testing; Cancer of Unknown Primary; CUP
MeSH Terms: conditions — Neoplasms, Unknown Primary; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Class 1, 2, or 3 alterations, with targeted therapy: Patients put on targeted therapies matched to specific genomic alterations.
- Site-specific therapy determined by tissue of origin testing: Patients put on therapy determined by tissue of origin testing (e.g., CancerTYPE ID)
- Empiric CUP therapy: Patients put on empiric treatment at physician discretion

SUMMARY:
The goal of the current study is to determine whether Foundation Medicine's next generation sequencing assay, called FoundationOne, will provide information that allows physicians to make treatment decisions using targeted therapies in clinical trials or FDA approved therapies, including "off-label" agents, that result in superior OS compared to historical outcomes for standard CUP therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histologically or cytologically confirmed diagnosis of metastatic or advanced unresectable cancer of unknown primary including adenocarcinoma, poorly differentiated adenocarcinoma, poorly differentiated carcinoma, or squamous carcinoma.
2. To be categorized as CUP, the following clinical evaluations must have been performed without identification of an anatomic primary site: medical history, physical examination, chemistry profile, blood counts, serum PSA (men), CT scans of chest/abdomen/pelvis, specific evaluation of symptomatic areas.
3. Sufficient Formalin Fixed Paraffin Embedded tissue from cancer of study will allow previously completed profiling panels other than for treatment assignment; however, FoundationOne profiling is required as part of this study. Adequate tumor tissue must remain, in the estimate of the consenting physician, to confirm genomic alterations in enrolled patients. Previous unknown primary available for FoundationOne testing. (Note: This FoundationOne® profiling is also allowed and is not required to be FoundationOne repeated.) (see Appendix A and Appendix B)
4. First and second line patients enrolling in this study must have an Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 to 2. Third line patients enrolling in this study must have an ECOG Performance Status score of 0 to 1 (Appendix C).
5. Patients must have measurable or evaluable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (Appendix D).
6. Age greater than or equal to 18 years.
7. Patients are considered potential candidates for treatment with targeted therapy.
8. Willingness and ability to comply with study and follow-up procedures.
9. Ability to understand the nature of this study and give written informed consent.
10. The presence of other active cancers is not allowed, unless indolent and not requiring therapy. Patients with early stage cancer who have received definitive local treatment and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e., non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.

Exclusion Criteria:

1. Patients who have received three or more lines of systemic therapy for cancer of unknown primary.
2. Patients who have previously received matched targeted therapy for the same Class 1 alteration (see Table 1) or the same drug.
3. Patients with treatable CUP syndrome, including the following:

   * extragonadal germ cell syndrome
   * neuroendocrine carcinoma
   * adenocarcinoma isolated to axillary lymph nodes (women)
   * peritoneal carcinomatosis (women)
   * squamous cell carcinoma limited to cervical, supraclavicular, or inguinal lymph nodes
   * single resectable metastasis
4. Previously untreated brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if therapy was completed at least 2 weeks prior to study entry and there is no evidence of central nervous system disease progression, mild neurologic symptoms, and no requirement for chronic corticosteroid therapy. Enzyme-inducing anticonvulsants are contraindicated.
5. Pregnant or lactating.
6. Psychological, familial, sociologic, or geographic conditions that do not permit compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed and previously treated patients with CUP.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2015-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Proportion of CUP patients who receive matched targeted therapy. | Baseline visit

SECONDARY OUTCOMES:
Overall survival (OS) in CUP patients receiving matched targeted therapy based on FoundationOne versus internal control CUP patients not receiving FoundationOne-directed therapy | Every three months until death, [20 months]

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation Medicine, Inc, Cambridge, Massachusetts, United States

REFERENCES:
- [Background] Drilon A, Wang L, Arcila ME, Balasubramanian S, Greenbowe JR, Ross JS, Stephens P, Lipson D, Miller VA, Kris MG, Ladanyi M, Rizvi NA. Broad, Hybrid Capture-Based Next-Generation Sequencing Identifies Actionable Genomic Alterations in Lung Adenocarcinomas Otherwise Negative for Such Alterations by Other Genomic Testing Approaches. Clin Cancer Res. 2015 Aug 15;21(16):3631-9. doi: 10.1158/1078-0432.CCR-14-2683. Epub 2015 Jan 7. PMID 25567908
- [Background] Ross JS, Cronin M. Whole cancer genome sequencing by next-generation methods. Am J Clin Pathol. 2011 Oct;136(4):527-39. doi: 10.1309/AJCPR1SVT1VHUGXW. PMID 21917674
- [Background] Frampton GM, Fichtenholtz A, Otto GA, Wang K, Downing SR, He J, Schnall-Levin M, White J, Sanford EM, An P, Sun J, Juhn F, Brennan K, Iwanik K, Maillet A, Buell J, White E, Zhao M, Balasubramanian S, Terzic S, Richards T, Banning V, Garcia L, Mahoney K, Zwirko Z, Donahue A, Beltran H, Mosquera JM, Rubin MA, Dogan S, Hedvat CV, Berger MF, Pusztai L, Lechner M, Boshoff C, Jarosz M, Vietz C, Parker A, Miller VA, Ross JS, Curran J, Cronin MT, Stephens PJ, Lipson D, Yelensky R. Development and validation of a clinical cancer genomic profiling test based on massively parallel DNA sequencing. Nat Biotechnol. 2013 Nov;31(11):1023-31. doi: 10.1038/nbt.2696. Epub 2013 Oct 20. PMID 24142049
- [Background] Johnson DB, Dahlman KH, Knol J, Gilbert J, Puzanov I, Means-Powell J, Balko JM, Lovly CM, Murphy BA, Goff LW, Abramson VG, Crispens MA, Mayer IA, Berlin JD, Horn L, Keedy VL, Reddy NM, Arteaga CL, Sosman JA, Pao W. Enabling a genetically informed approach to cancer medicine: a retrospective evaluation of the impact of comprehensive tumor profiling using a targeted next-generation sequencing panel. Oncologist. 2014 Jun;19(6):616-22. doi: 10.1634/theoncologist.2014-0011. Epub 2014 May 5. PMID 24797823
- [Background] Tsimberidou AM, Iskander NG, Hong DS, Wheler JJ, Falchook GS, Fu S, Piha-Paul S, Naing A, Janku F, Luthra R, Ye Y, Wen S, Berry D, Kurzrock R. Personalized medicine in a phase I clinical trials program: the MD Anderson Cancer Center initiative. Clin Cancer Res. 2012 Nov 15;18(22):6373-83. doi: 10.1158/1078-0432.CCR-12-1627. Epub 2012 Sep 10. PMID 22966018
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Massard C, Loriot Y, Fizazi K. Carcinomas of an unknown primary origin--diagnosis and treatment. Nat Rev Clin Oncol. 2011 Nov 1;8(12):701-10. doi: 10.1038/nrclinonc.2011.158. PMID 22048624
- [Background] Pavlidis N, Pentheroudakis G. Cancer of unknown primary site. Lancet. 2012 Apr 14;379(9824):1428-35. doi: 10.1016/S0140-6736(11)61178-1. Epub 2012 Mar 12. PMID 22414598
- [Background] Stella GM, Senetta R, Cassenti A, Ronco M, Cassoni P. Cancers of unknown primary origin: current perspectives and future therapeutic strategies. J Transl Med. 2012 Jan 24;10:12. doi: 10.1186/1479-5876-10-12. PMID 22272606
- [Background] Gray SW, Hicks-Courant K, Cronin A, Rollins BJ, Weeks JC. Physicians' attitudes about multiplex tumor genomic testing. J Clin Oncol. 2014 May 1;32(13):1317-23. doi: 10.1200/JCO.2013.52.4298. Epub 2014 Mar 24. PMID 24663044
- [Background] Varadhachary GR, Raber MN. Carcinoma of unknown primary site. N Engl J Med. 2014 Nov 20;371(21):2040. doi: 10.1056/NEJMc1411384. No abstract available. PMID 25409386
- [Background] Petrakis D, Pentheroudakis G, Voulgaris E, Pavlidis N. Prognostication in cancer of unknown primary (CUP): development of a prognostic algorithm in 311 cases and review of the literature. Cancer Treat Rev. 2013 Nov;39(7):701-8. doi: 10.1016/j.ctrv.2013.03.001. Epub 2013 Apr 6. PMID 23566573
- [Background] Hainsworth JD, Rubin MS, Spigel DR, Boccia RV, Raby S, Quinn R, Greco FA. Molecular gene expression profiling to predict the tissue of origin and direct site-specific therapy in patients with carcinoma of unknown primary site: a prospective trial of the Sarah Cannon research institute. J Clin Oncol. 2013 Jan 10;31(2):217-23. doi: 10.1200/JCO.2012.43.3755. Epub 2012 Oct 1. PMID 23032625
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009